CLINICAL TRIAL: NCT00681525
Title: A Multiple-Dose Pharmacokinetic Interaction Study Between ABT-335, Atorvastatin and Ezetimibe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Maureen Kelly, MD, Abbott
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M10-367
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-09

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; fenofibric acid; Atorvastatin; Ezetimibe

ARMS (3):
- A (Experimental): ABT-335 135 mg
  Interventions: Drug: ABT-335
- B (Experimental): Atorvastatin 80 mg and Ezetimibe 10 mg
  Interventions: Drug: Atorvastatin; Drug: Ezetimibe
- C (Experimental): ABT-335 135 mg, Atorvastatin 80 mg and Ezetimibe 10 mg
  Interventions: Drug: ABT-335; Drug: Atorvastatin; Drug: Ezetimibe

INTERVENTIONS:
Drug: ABT-335 — One ABT-335 135 mg capsule QD for 10 days
  Other Names: fenofibric acid
  Arms: A; C
Drug: Atorvastatin — One 80 mg tablet of atorvastatin QD for 10 days
  Other Names: atovastatin
  Arms: B; C
Drug: Ezetimibe — One ezetimibe 10 mg tablet QD for 10 days
  Arms: B; C

SUMMARY:
The objective of this study is to evaluate the potential PK interaction between ABT-335, atorvastatin 80 mg and ezetimibe 10 mg when administered concurrently.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects

Exclusion Criteria:

* Clinically significant diseases or disorders
* Positive screens for drug and alcohol
* Pregnant or breast-feeding females
* Any history of surgery(ies) that might interfere with the gastrointestinal motility, pH or absorption

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
PK interaction | Study duration approximately 62 days

CONTACTS AND LOCATIONS:
Locations (1):
- Site Reference ID/Investigator# 8087, Gainesville, Florida, United States